CLINICAL TRIAL: NCT04091854
Title: A Study to Observe the Progress of Diabetes Mellitus After 52 or 28 Weeks of HMS5552 Treatment for Type 2 Diabetes Mellitus
Brief Title: The Progress of Diabetes Mellitus After HMS5552 Treatment in Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Majianhua (Other)
Responsible Party: Sponsor-Investigator, Majianhua, Director, Head of Endocrinology department, Clinical Professor, Nanjing First Hospital, Nanjing Medical University
Organization: Nanjing First Hospital, Nanjing Medical University (Other)
Other Study IDs: KY20190530-01-KS-01
Record Dates: First submitted 2019-09-01; First posted 2019-09-17 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2020-12

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Glucokinase Activator; Glucose control
MeSH Terms: interventions — Dorzagliatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HMS5552 treatment
  Interventions: Drug: HMS5552

INTERVENTIONS:
Drug: HMS5552 — To observe the progress of diabetes mellitus after 52 or 28 weeks of HMS5552 treatment for type 2 diabetes mellitus

SUMMARY:
At present, there are few studies on the clinical remission rate of diabetes after one year discontinuation of oral hypoglycemic drugs after intensive treatment. HMS5552 is a kind of GKA hypoglycemic drug. This study intends to observe the clinical remission rate of diabetes mellitus, beta cell function and blood sugar fluctuation of patients with type 2 diabetes mellitus who have been treated with HMS5552 for 52W or 28W and whose glucose control is up to the standard.

ELIGIBILITY:
Inclusion Criteria:

* Complete HMS5552 treatment and safety visit;
* HbA1c < 8.0% was detected in our laboratory;
* Researchers judged the stability of glucose control based on the data of subjects'visits during HMS5552 treatment and the indicators of our hospital;
* Subjects are able and willing to monitor peripheral blood sugar and regularity of diet and exercise;
* Willing to sign written informed consent and abide by the research program.

Exclusion Criteria:

* There was a state of illness in the subjects who could not complete the follow-up during the observation period.
* The researchers judged that subjects'compliance with HMS5552 was affected during treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, subjects with type 2 diabetes mellitus treated with HMS5552 were screened to meet the target of glucose control when they completed 52 or 28 weeks of HMS5552 treatment respectively.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 4 weeks
  Changes of HbA1c
Fasting glucose | 4 weeks
  Changes of fasting glucose
Postprandial glucose | 4 weeks
  Changes of postprandial glucose
C peptide | 4-8 weeks
  Changes of C peptide

SECONDARY OUTCOMES:
TNF-α | 52 weeks
  Changes of TNF-α
IL-6 | 52 weeks
  Changes of IL-6
8-iso PGF2α | 52 weeks
  Changes of 8-iso PGF2α

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided